CLINICAL TRIAL: NCT06270173
Title: A Prospective, Multicenter, Open-Label, Post-Market Study to Evaluate The Effectiveness and Safety of The Tripod-Fix Vertebral Body Augmentation System in Osteoporotic Vertebral Compression Fractures Treatment
Brief Title: Post-Market Study of The Tripod-Fix Vertebral Body Augmentation System in Osteoporotic Vertebral Compression Fractures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wiltrom Co., Ltd. (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TWM-C-2202
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Osteoporotic Vertebral Compression Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Tripod-Fix will be used to treat osteoporotic vertebral compression fractures.
  Interventions: Device: Tripod-Fix Vertebral Body Augmentation System (Tripod-Fix)

INTERVENTIONS:
Device: Tripod-Fix Vertebral Body Augmentation System (Tripod-Fix) — The Tripod-Fix is a permanent implant used for vertebral augmentation in patients with osteoporotic vertebral compression fractures.

SUMMARY:
The objective of this Post-Market Clinical Follow-Up Study is to evaluate the safety and performance of the Tripod-Fix in the treatment of vertebral compression fractures (VCF) resulting from osteoporosis.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label, single-arm, PMCF study. The sample size for this study will be 50 patients. Eligible patients will be treated with Tripod-Fix on Day 0 and will be followed for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form prior to any study procedures
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Skeletally mature males and females
4. 1 painful VCF which meets all of the following criteria:

   1. Fracture due to diagnosed or presumed underlying osteoporosis (T-score < -2.5 points)
   2. VCF between T6 and L5
   3. VCF shows loss of height in the anterior, mid or posterior third of the vertebral body from an estimated pre-fracture configuration, but no more than 50% based on X-ray, CT or MRI at baseline.
   4. The Index fracture is acute or persistent (not healed), as demonstrated by MRI (or bone scan if the patient is contraindicated for MRI).
5. Investigator believes target vertebral body is suitable for Tripod-Fix procedure (e.g., appropriate pedicle diameter) assessed on radiography preoperative.

Exclusion Criteria:

Tripod-Fix is not indicated for any other application other than that for which it is designed. contraindications for Tripod-Fix include, but are not limited to: .

1. Patient presenting a loss of vertebral height >50% compared to estimated pre-fracture height
2. Sclerotic fracture
3. Patient with a prior history of intolerance or of allergic reaction to titanium and/or one of the components of the PMMA cement
4. Patient suffering from irreversible coagulopathy or undergoing anticoagulant treatment at the moment of surgery or at least 8 days prior to inclusion
5. Active infection (systemic or in the target vertebra)
6. Patient suffering from a severe or uncontrolled systemic disease
7. Patient presenting a pathological fracture with the presence of a mass within the spinal canal
8. Patient presenting neurological damage caused by vertebral fracture
9. Patient pregnant or likely to be so or breastfeeding
10. Patient vertebral anatomy not compatible with the size of the implant or instrumentation
11. Fracture geometry making the insertion of the implant impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with study success | 12 months post-procedure
  Study success is defined as follows:
  1. The reduction of Visual Analogue Scale (VAS) score > 20 mm at the 12 month follow up visit compared to baseline as measured by the 100-mm VAS measurement, AND
  2. Maintenance or improvement in function at the 12 month follow up visit compared to baseline as measured by the 100-point Oswestry Disability Index (ODI) AND,
  3. Absence of device-related serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Te-Yang Tsai, Study Director — Wiltrom Co., Ltd.
Locations (4):
- Germany (4):
  - Klinikum Friedrichshafen, Friedrichshafen, Baden-Wurttemberg
  - University Hospital Mannheim, Mannheim, Baden-Wurttemberg
  - Johann Wolfgang Goethe University Frankfurt/Main, Frankfurt am Main, Hesse
  - Krankenaus Mechernich, Mechernich, North Rhine-Westphalia